CLINICAL TRIAL: NCT07185542
Title: Function-Preserving Surgery for Parotid Tumors: Intracapsular Versus Superficial Parotidectomy; A Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sayed Abd El Bary, Prinicipal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Parotid Tumors Surgery
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parotid Tumors; Parotidectomy
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracapsular parotidectomy (Active Comparator): ICP is recommended for small, mobile, and superficially located benign tumors with low suspicion of malignancy. However, concerns remain regarding capsular rupture and recurrence, particularly in pleomorphic adenomas with microscopic extensions
  Interventions: Procedure: Intracapsular parotidectomy (ICP)
- Superficial parotidectomy (Active Comparator): Superficial parotidectomy (SP), the traditional approach, involves facial nerve dissection and removal of the superficial lobe. Though effective, it carries risks like nerve dysfunction, Frey's syndrome, and cosmetic concerns
  Interventions: Procedure: Superficial parotidectomy

INTERVENTIONS:
Procedure: Superficial parotidectomy — Superficial parotidectomy (SP), the traditional approach, involves facial nerve dissection and removal of the superficial lobe. Though effective, it carries risks like nerve dysfunction, Frey's syndrome, and cosmetic concerns
  Arms: Superficial parotidectomy
Procedure: Intracapsular parotidectomy (ICP) — ICP excises the tumor along its capsule without dissecting the facial nerve, thereby minimizing trauma and preserving glandular tissue.
  ICP is recommended for small, mobile, and superficially located benign tumors with low suspicion of malignancy. However, concerns remain regarding capsular rupture and recurrence, particularly in pleomorphic adenomas with microscopic extensions
  Arms: Intracapsular parotidectomy

SUMMARY:
Benign parotid gland tumors, such as pleomorphic adenoma and Warthin tumors, constitute the majority of salivary gland neoplasms. Surgical excision remains the primary treatment, traditionally achieved through superficial parotidectomy (SP). However, SP may lead to complications such as facial nerve dysfunction, Frey's syndrome, and aesthetic concerns. Intracapsular parotidectomy (ICP), a minimally invasive alternative, aims to minimize surgical morbidity while preserving oncologic safety. This study aimes to compare intracapsular parotidectomy and superficial parotidectomy in terms of operative efficiency, complications, facial nerve preservation, and tumor recurrence for benign parotid tumors.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 65 years,
* radiologically and clinically confirmed benign parotid tumor
* tumor confined to the superficial or deep lobe without evidence of facial nerve involvement.

Exclusion Criteria:

* suspicion of malignancy based on imaging or fine-needle aspiration cytology (FNAC)
* recurrent parotid tumors
* previous parotid surgery
* facial nerve dysfunction preoperatively
* comorbidities precluding surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperatively
Blood Loss | Introperative
  Measuring the amount of blood loss introperatively
recurrence rate | 6 months postopeartively

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Madīnat an Naşr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided